CLINICAL TRIAL: NCT01691729
Title: A Randomized, Multicenter, Cross-Over Study Comparing the Performance of Three Ostomy Accessory Products
Brief Title: Comparison Study of 3 Ostomy Products
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ConvaTec Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A739
Record Dates: First submitted 2012-09-12; First posted 2012-09-25 (Estimated); Last update posted 2022-12-07 (Actual); Status verified 2022-12

CONDITIONS: Ostomy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (6):
- Ostomy 1 (Other): 3 Ostomy Accessory Devices with the order of wear being Investigative Ostomy AccessoryProduct/Ostomy Accessory Marketed Product #1/Ostomy Accessory Marketed Product #2
  Interventions: Device: Ostomy accessory
- Ostomy 2 (Other): 3 Ostomy Accessory Devices with the order of wear being Investigative Ostomy Accessory Product/Ostomy Accessory Marketed Product #2/Ostomy Accessory Marketed Product #1
  Interventions: Device: Ostomy accessory
- Ostomy 3 (Other): 3 Ostomy Accessory Devices with the order of wear being Ostomy Accessory Marketed Product #1/Ostomy Accessory Marketed Product #2/Investigative Ostomy Accessory Product
  Interventions: Device: Ostomy accessory
- Ostomy 4 (Other): 3 Ostomy Accessory Devices with the order of wear being Ostomy Accessory Marketed Product #2/Ostomy Accessory Marketed Product #1/Investigative Ostomy Accessory Product
  Interventions: Device: Ostomy accessory
- Ostomy 5 (Other): 3 Ostomy Accessory Devices with the order of wear being Ostomy Accessory Marketed Product #1/Investigative Ostomy Accessory Product/Ostomy Accessory Marketed Product #2
  Interventions: Device: Ostomy accessory
- Ostomy 6 (Other): 3 Ostomy Accessory Devices with the order of wear being Ostomy Accessory Marketed Product #2/Investigative Ostomy Accessory Product/Ostomy Accessory Marketed Product #1
  Interventions: Device: Ostomy accessory

INTERVENTIONS:
Device: Ostomy accessory — Wearing each of the devices for 10 days each

SUMMARY:
To purpose of the study is to evaluate and compare the efficacy of three ostomy accessory products.

DETAILED DESCRIPTION:
The primary objective of this study was to evaluate and compare the efficacy of three ostomy accessory products in terms of leakage and wear time. Secondary objectives were to evaluate and compare the safety of three ostomy accessory products, and to assess and compare the performance of the three products in terms of use and overall impression.

ELIGIBILITY:
Inclusion Criteria:

* Has an ostomy
* Is at least 18 years of age
* Has a stoma for at least 3 months
* Other than thier ostomy is considered to have a healthy/stable health
* Is able to take care of their stoma

Exclusion Criteria:

* Known sensitivity to any of the ostomy devices or components
* Is undergoing chemotherapy or radiotherapy
* Has participated in a clinical study within the past 30 days
* Has a medical condition, in which in the opinion of the Investigator would not be a good candidate for the study and justifies exclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Leakage & Wear Time | 10 days
  Evaluation and comparison of the efficacy of three ostomy accessory products in terms of leakage and wear time.

SECONDARY OUTCOMES:
Number of adverse events | 10 days
  Evaluation and comparison of the safety of three ostomy accessory products

CONTACTS AND LOCATIONS:
Overall Officials: Kim Peters, Study Director — ConvaTec Inc.
Locations (4):
- United States (4):
  - Independent Nurse Consultants, Tucson, Arizona
  - ET Nursing Services, Jacksonville, Florida
  - Image Specialties, Saint Joseph, Missouri
  - ID MED Inc., Columbus, Ohio